CLINICAL TRIAL: NCT01494194
Title: Evaluation of the Potential of Air Structuring Protein, a Novel Protein Preparation Derived From Trichoderma Reesei, to Elicit Allergic Reactions in Mold Sensitized People
Brief Title: Study to Evaluate the Potential of Air Structuring Protein to Elicit Allergic Reactions in Mold Sensitized People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever SEAC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: KQC100140
Record Dates: First submitted 2011-12-12; First posted 2011-12-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Allergy to Mold
Keywords: Mold sensitized

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo for food challenge (Placebo Comparator)
  Interventions: Other: Placebo sorbet
- ASP Skin prick solution (Experimental)
  Interventions: Other: Air Structuring Protein
- ASP sorbet (Experimental)
  Interventions: Other: Air Structuring Protein

INTERVENTIONS:
Other: Air Structuring Protein — A novel food protein preparation
  Arms: ASP Skin prick solution; ASP sorbet
Other: Placebo sorbet — Placebo sorbet for double blind placebo controlled food challenge
  Arms: placebo for food challenge

SUMMARY:
Air Structuring Protein (ASP) is a small protein derived from a fungus which is already widely used to produce enzymes that are added to foods. ASP has the possibility of stabilising the air phase of ice-cream and therefore there is interest in ASP as a potential ice-cream ingredient.

Toxicological tests have also been carried out to further confirm the safety of the material and no evidence of genotoxicity or acute toxicity has been observed in any of the tests.

As part of the safety evaluation of a new protein for use in foods, the potential allergenicity is also investigated and Unilever is sponsoring a study to evaluate this aspect of ASP. This study will investigate:

* Whether ASP has the potential to elicit a positive skin prick test (SPT) in a population of participants with proven sensitivity to mould.
* Whether ASP is responsible for any positive SPT reactions, should they occur.
* And if any positive SPT reactions to ASP occur, whether such reactions are clinically relevant with respect to food allergy.

The study is divided in three stages. In Stage 1 and Stage 2, the SPT is "open label," which means that both the participant and the study doctor will know which materials are being tested.

In Stage 3, the food challenge has a "crossover" design, meaning that participants will take one of the products (ASP or placebo [food containing no ASP]) during the first half of the study and the other treatment during the second half. The order of ASP and placebo will be decided randomly, like tossing a coin. To make the comparison between ASP and placebo as fair as possible, the food challenge is "double blinded." This means that neither the participant nor the study doctor will know which kind of products (ASP or placebo) the participant is taking.

This is a multi centre study which is taking place in the UK.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-60 years.
* Mould sensitised subjects diagnosed according to the EAACI/Ga2len guidelines.
* Written informed consent from the subject.
* Normally active and otherwise judged to be in good health on the basis of medical history and screening assessment.
* No allergic symptoms on the day of investigation.

Exclusion Criteria:

* Pregnancy or lactation.
* Failure to comply with the protocol.
* Medication that may interfere with wheal formation in the skin or response to DBPCFC
* Participation in another clinical study involving a SPT within 30 days prior to Visit 1 or DBPCFC within 30 days prior to DBPCFC.
* Current skin disease of any type (eczema, acne, dermatitis, etc.) on the test site(s).
* Subjects with a condition the Investigator believes would interfere with the evaluation of the subject, including proceeding to DBPCFC, or may put the subject at undue risk, e.g., a history of anaphylactic reactions and history of reactions to any component of the DBPCFC matrix other than ASP.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Positive skin prick test response to test material | 15 minutes after application
  The number and size of positive SPTs will be recorded together with data of concomitant allergies and the minimum eliciting concentration (SPT-min) in the skin.

SECONDARY OUTCOMES:
The number of positive Double Blind Placebo Controlled Food Challenge reactions in those with positive skin prick test result | 2 hours after administration
  The number of positive DBPCFC reactions will be recorded together with pre and post challenge blood pressure, pulse rate, peak expiratory flow (PEF) and forced expiratory volume (FEV1), data of concomitant allergies, any symptoms elicited including any late onset reactions, timing of symptoms and the minimum eliciting dose of ASP.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart and Lung Institute, MRC & Asthma UK Centre in Allergic Mechanisms of Asthma, Centre for Respiratory Infection, Imperial College London, London, United Kingdom